CLINICAL TRIAL: NCT04922320
Title: Effect of Patient Priorities Care Implementation in Older Veterans With Multiple Chronic Conditions
Acronym: PPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 20-079; 1 I01 HX003211-01A1 (Other Grant/Funding Number: VA Office of Research and Development); CIN 13-413 (Other Grant/Funding Number: VA IQuESt Center)
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Multiple Chronic Conditions; Decision Making, Shared
Keywords: Patient Centered Care; Geriatrics
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: All consented participants who complete baseline assessment will be randomized into the PPC or UC groups. Randomization will be blocked and stratified by PCP to assure balance in the number of patients assigned to two study arms by enrolled PCP. Within each clinician, the investigators will use random blocks of 4 and 6. Blocking ensures half will be randomized to PPC and half to UC. Varying block size makes the sequence of assignments more difficult to predict. The random numbers will be generated in SAS PROC PLAN. The research assistant (RA) conducting baseline evaluations will not access any randomization procedures, leaving that RA blinded during the evaluation.
Who Masked: Outcomes Assessor
Masking Description: The research assistant (RA) conducting baseline evaluations will not access any randomization procedures, leaving that RA blinded during the evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Priorities Care (Experimental): A facilitator will schedule a PPC facilitation encounter 2-3 weeks before an upcoming PCP visit. The facilitator conducts a structured assessment using a written conversation guide that begins with general questions establishing what is most important to Veterans about their health and moves toward establishing specific goals (actionable outcomes), and what patients are willing/not willing to do to achieve these goals (care preferences). The result is a structured patient priorities report delivered to PCPs designed to facilitate changes in the patient's care plan to align it with his/her priorities. In the subsequent visit, the PCP will use one or more of the established PPC decisional strategies to align care with patients' priorities. Education for PCPs about the facilitation process, the patient priorities report, and the decisional strategies occurs prior to the PCP seeing any intervention patients. The PCP will document changes in care made to achieve the identified priorities.
  Interventions: Behavioral: Patient Priorities Care
- Usual Care (Placebo Comparator): PCPs will not be alerted when an encounter involves a UC group participant. UC participant visits will appear the same as all other unenrolled patient encounters. UC participants will not receive any additional preparation
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Patient Priorities Care — A facilitator will schedule a PPC facilitation encounter 2-3 weeks before an upcoming PCP visit. The facilitator conducts a structured assessment using a written conversation guide that begins with general questions establishing what is most important to Veterans about their health and moves toward establishing specific goals (actionable outcomes), and what patients are willing/not willing to do to achieve these goals (care preferences). The result is a structured patient priorities report delivered to PCPs designed to facilitate changes in the patient's care plan to align it with his/her priorities. In the subsequent visit, the PCP will use one or more of the established PPC decisional strategies to align care with patients' priorities. Education for PCPs about the facilitation process, the patient priorities report, and the decisional strategies occurs prior to the PCP seeing any intervention patients. The PCP will document changes in care made to achieve the identified priorities.
  Arms: Patient Priorities Care
Other: Usual Care — PCPs will not be alerted when an encounter involves a UC group participant. UC participant visits will appear the same as all other unenrolled patient encounters. PCPs will be trained to address the needs of UC participants based on their typical approach without the use of a facilitator or explicit process for identifying patient priorities. UC participants will not receive any additional preparation
  Arms: Usual Care

SUMMARY:
The investigators will conduct a randomized control trial enrolling 420 older Veterans with multiple chronic conditions receiving primary care at the Michael E. DeBakey VA Medical Center and VA Connecticut Medical Center to determine if Patient Priorities Care reduces treatment burden, increases priorities-aligned home and community services, and sets shared health outcome goals compared with usual care. The investigators will randomize at the patient level rather than clinic or clinician level to evaluate the effect of identifying patient priorities on clinician decision making and alignment of care with identified priorities.

ELIGIBILITY:
Inclusion Criteria:

* 2 encounters in prior 18 months
* 3 active health problems on active problem list or prescribed 10 medications

Exclusion Criteria:

* nursing home resident
* end stage renal disease on dialysis
* active serious mental illness (psychosis, schizophrenia, etc)
* active substance use disorder
* complete hearing loss
* dementia
* Non-English speaker (translator required)
* 4 or more no-show appointments in the last 6 months
* the investigators will present a list of eligible patients to PCPs prior to chart review to identify patients who the PCP:

  * a) believes cannot participate independently or provide informed consent due to cognitive impairment
  * b) "would not be surprised if the patient passed away within the next 12 months?"

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 420 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Reported Treatment Burden | 4 month follow-up
  Measured by the validated Treatment Burden Questionnaire, treatment burden measures perceptions of burdensomeness of overall care and treatment burden (e.g., medication taking, self-monitoring, visits to the provider, tests, tasks to access and coordinate care) imposed by healthcare as assessed with 15 items; possible range, 0-150; Cronbach = 0.90; higher scores indicate greater perceived burden.
Home and Community Services Use | 4 month follow-up
  Home and community based services includes care that supports independence and the ability to stay in one's own home. They are defined by the VA Geriatrics and Extended Care Data Analysis Center (GEC-DAC) as VA Long Term Services and Supports: adult day health care, home based primary care, homemaker and home health aide, hospice care, palliative care, respite care, skilled home health care, home telehealth, and home care services. GEC-DAC has created a composite measure, which is associated with delays in nursing home and institutional long-term care placement.

SECONDARY OUTCOMES:
shared decision making | 4 month follow-up
  Measured using the CollaboRATE scale (3 items; possible range 0-100; Cronbach = 0.89; higher score indicates greater perceived shared decision-making and goal ascertainment).
Patients' goal setting | 4 month follow-up
  Will measure patients' perceptions of whether health care decisions were collaborative and focused on their goals using the Older Patient Assessment of Chronic Illness Care (OPACIC) score (11 items; range, 1-5; Cronbach = 0.87; higher scores indicate better perceived chronic disease care).
Ambulatory Care Utilization | 4 month follow-up
  Medications added or stopped and diagnostic tests, referrals, and procedures ordered or avoided. Measured using a structured chart review tool using our validated process to guide uniform abstraction and classification to a) document specific changes in treatment (i.e., medications, referrals, diagnostics, self-care, services and supports), b) attribute changes to alignment with priorities, and c) identify documentation of any avoided care.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian N. Dindo, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen AB, Paiva AL, Redding CA, Fried TR. Characteristics of Older Adults Who Cannot Identify a Healthcare Agent. J Gen Intern Med. 2022 Apr;37(5):1313-1314. doi: 10.1007/s11606-021-06798-2. Epub 2021 Apr 26. No abstract available. PMID 33904034
- [Background] Ouellet GM, Fried TR, Gilstrap LG, O'Leary JR, Austin AM, Skinner JS, Cohen AB. Anticoagulant Use for Atrial Fibrillation Among Persons With Advanced Dementia at the End of Life. JAMA Intern Med. 2021 Aug 1;181(8):1121-1123. doi: 10.1001/jamainternmed.2021.1819. PMID 33970197
- [Result] Vaughan EM, Johnson E, Naik AD, Amspoker AB, Balasubramanyam A, Virani SS, Ballantyne CM, Johnston CA, Foreyt JP. Long-Term Effectiveness of the TIME Intervention to Improve Diabetes Outcomes in Low-Income Settings: a 2-Year Follow-Up. J Gen Intern Med. 2022 Sep;37(12):3062-3069. doi: 10.1007/s11606-021-07363-7. Epub 2022 Feb 7. PMID 35132555
- [Result] Naik AD, Walling AM. Getting patients ready for "in the moment" decisions. J Am Geriatr Soc. 2022 Sep;70(9):2474-2477. doi: 10.1111/jgs.17935. Epub 2022 Jul 4. No abstract available. PMID 35781226
- [Result] Lee YK, Fried TR, Costello DM, Hajduk AM, O'Leary JR, Cohen AB. Perceived dementia risk and advance care planning among older adults. J Am Geriatr Soc. 2022 May;70(5):1481-1486. doi: 10.1111/jgs.17721. Epub 2022 Mar 11. PMID 35274737
- [Result] Zang E, Shi Y, Wang X, Wu B, Fried TR. Trajectories of physical functioning among US adults with cognitive impairment. Age Ageing. 2022 Jun 1;51(6):afac139. doi: 10.1093/ageing/afac139. PMID 35751871
- [Result] Fried TR. Giving up on the objective of providing goal-concordant care: Advance care planning for improving caregiver outcomes. J Am Geriatr Soc. 2022 Oct;70(10):3006-3011. doi: 10.1111/jgs.18000. Epub 2022 Aug 16. PMID 35974460
- [Result] Amenta E, Grigoryan L, Rajan SS, Ramsey D, Kramer JR, Walder A, Chou A, Van JN, Krein SL, Hysong S, Naik AD, Trautner BW. Quantifying the Implementation and Cost of a Multisite Antibiotic Stewardship Intervention for Asymptomatic Bacteriuria. Antimicrob Steward Healthc Epidemiol. 2023 Jun 30;3(1):e115. doi: 10.1017/ash.2023.198. eCollection 2023. PMID 37502251
- [Result] Dindo L, Chaison A, Rodrigues M, Woods K, Mark A, Boykin D. Feasibility of delivering a virtual 1-day acceptance and commitment therapy workshop to rural veterans through community partnerships. Contemp Clin Trials Commun. 2023 Jun 20;34:101178. doi: 10.1016/j.conctc.2023.101178. eCollection 2023 Aug. PMID 37409189
- [Result] Chary AN, Brickhouse E, Torres B, Santangelo I, Carpenter CR, Liu SW, Godwin KM, Naik AD, Singh H, Kennedy M. Leveraging the Electronic Health Record to Implement Emergency Department Delirium Screening. Appl Clin Inform. 2023 May;14(3):478-486. doi: 10.1055/a-2073-3736. Epub 2023 Apr 13. PMID 37054983
- [Result] Chary A, Brickhouse E, Torres B, Cameron-Comasco L, Lee S, Punches B, Skains RM, Naik AD, Quatman-Yates CC, Kennedy M, Southerland LT, Liu S. Physical therapy consultation in the emergency department for older adults with falls: A qualitative study. J Am Coll Emerg Physicians Open. 2023 Apr 19;4(2):e12941. doi: 10.1002/emp2.12941. eCollection 2023 Apr. PMID 37090953
- [Result] Chary A, Hernandez N, Rivera AP, Ramont V, Obi T, Santangelo I, Ritchie C, Singh H, Hayden E, Naik AD, Liu S, Kennedy M. Perceptions of Acute Care Telemedicine Among Caregivers for Persons Living with Dementia: A Qualitative Study. J Appl Gerontol. 2024 Jan;43(1):69-77. doi: 10.1177/07334648231198018. Epub 2023 Sep 8. PMID 37682526
- [Result] Freytag J, Mishra RK, Street RL Jr, Catic A, Dindo L, Kiefer L, Najafi B, Naik AD. Using Wearable Sensors to Measure Goal Achievement in Older Veterans with Dementia. Sensors (Basel). 2022 Dec 16;22(24):9923. doi: 10.3390/s22249923. PMID 36560290
- [Result] Razjouyan J, Horstman MJ, Orkaby AR, Virani SS, Intrator O, Goyal P, Amos CI, Naik AD. Developing a Parsimonious Frailty Index for Older, Multimorbid Adults With Heart Failure Using Machine Learning. Am J Cardiol. 2023 Mar 1;190:75-81. doi: 10.1016/j.amjcard.2022.11.044. Epub 2022 Dec 23. PMID 36566620
- [Result] Crespo-Ramos G, Bebu I, Krause-Steinrauf H, Hoogendoorn CJ, Fang R, Ehrmann D, Presley C, Naik AD, Katona A, Walker EA, Cherrington A, Gonzalez JS; GRADE Research Group. Emotional distress and cardiovascular disease risk among participants enrolled in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness (GRADE) study. Diabetes Res Clin Pract. 2023 Sep;203:110808. doi: 10.1016/j.diabres.2023.110808. Epub 2023 Jun 30. PMID 37394014
- [Result] Ritchey KC, Solberg LM, Citty SW, Kiefer L, Martinez E, Gray C, Naik AD. Guiding Post-Hospital Recovery by 'What Matters:' Implementation of Patient Priorities Identification in a VA Community Living Center. Geriatrics (Basel). 2023 Jul 4;8(4):74. doi: 10.3390/geriatrics8040074. PMID 37489322
- [Result] Chary AN, Torres B, Brickhouse E, Santangelo I, Godwin KM, Naik AD, Carpenter CR, Liu SW, Kennedy M. Language discordance in emergency department delirium screening: Results from a qualitative interview-based study. J Am Geriatr Soc. 2023 Apr;71(4):1328-1331. doi: 10.1111/jgs.18147. Epub 2022 Nov 30. No abstract available. PMID 36451059
- [Result] Chary AN, Naik AD, Kennedy M. Reply to: Expanding options to include language barriers for predicting postoperative delirium in geriatric patients. J Am Geriatr Soc. 2023 Jan;71(1):294-295. doi: 10.1111/jgs.18083. Epub 2022 Oct 17. No abstract available. PMID 36254368
- [Result] Naik AD. Measuring patient-centered care to improve hospital experiences of older adults. J Am Geriatr Soc. 2022 Dec;70(12):3348-3351. doi: 10.1111/jgs.18048. Epub 2022 Sep 20. No abstract available. PMID 36125214
- [Result] Scholle SH, Naik AD. A Person-Centered Care Dashboard for Individuals With Complex Health Care Needs-Charting a Course for the Future. JAMA Netw Open. 2022 Aug 1;5(8):e2224945. doi: 10.1001/jamanetworkopen.2022.24945. No abstract available. PMID 35917127

DOCUMENTS (1):
  • Informed Consent Form (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT04922320/ICF_000.pdf